CLINICAL TRIAL: NCT00478595
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Assess the Efficacy and Safety of SR141716 in Obese Type 2 Diabetic Patients on Monotherapy Inadequately Controlled With Oral Anti-diabetic Drug
Brief Title: Japanese Study With Rimonabant in Obese Type 2 Diabetic Patients With Oral Anti-diabetic Drug
Acronym: SYMPHONY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision taken in light of demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC6647
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Obesity; Diabetes Mellitus Type 2
Keywords: obese; diabetes; cannabinoid-1 receptor
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rimonabant (Experimental): Rimonabant 20 mg once daily
  Interventions: Drug: Rimonabant; Drug: Anti-diabetic monotherapy
- Placebo (Placebo Comparator): Placebo (for Rimonabant) once daily
  Interventions: Drug: Placebo (for Rimonabant); Drug: Anti-diabetic monotherapy

INTERVENTIONS:
Drug: Rimonabant — Tablet, oral administration
  Other Names: SR141716; Acomplia
  Arms: Rimonabant
Drug: Placebo (for Rimonabant) — Tablet, oral administration
  Arms: Placebo
Drug: Anti-diabetic monotherapy — Previous treatment with Sulfonylurea or α-glucosidase inhibitor continued at stable dose during the study period

SUMMARY:
The primary objective of this study is to assess the efficacy of Rimonabant (SR141716) compared to placebo on change in HbA1c and on relative change in body weight over 52 weeks in obese type 2 diabetic patients on monotherapy inadequately controlled with oral anti-diabetic drug (sulfonylurea or α-glucosidase inhibitor).

The secondary objectives are:

* To evaluate the effect of Rimonabant compared to placebo on other parameters related to the glucose control, waist circumference, Body Mass Index and metabolic parameters;
* To evaluate the safety and tolerability of Rimonabant compared to placebo;
* To evaluate the pharmacokinetics of Rimonabant.

DETAILED DESCRIPTION:
The total duration per patient will be approximately 69 weeks including a 52-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus patients on monotherapy with oral anti-diabetic drug (sulfonylurea or α-glucosidase inhibitor)
* HbA1C ≥ 7.0 % and ≤ 10.0 %
* Body Mass Index ≥ 25 kg/m²

Exclusion Criteria:

* Type 1 diabetes
* Within 12 weeks prior to screening visit: use of oral antidiabetic drugs (other than a sulfonylurea or alpha-glucosidase inhibitor) and/or insulin, of anti-obesity drugs or other drugs for weight reduction
* Within 4 weeks prior to screening visit: administration of systemic long-acting corticosteroids or prolonged use (more than one week) of other systemic corticosteroids, change in lipid lowering treatment
* Secondary obesity
* Primary hyperlipidemia
* Positive serum pregnancy test in females of childbearing potential

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in HbA1C | Baseline to week 52
Relative change from baseline in in body weight | Baseline to week 52

SECONDARY OUTCOMES:
Absolute change from baseline in Fasting Plasma Glucose | Baseline to week 52
Absolute change from baseline in waist circumference | Baseline to week 52
Relative change from baseline in Triglycerides and HDL-cholesterol | Baseline to week 52
Safety: overview of adverse events | Baseline to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan